CLINICAL TRIAL: NCT06584864
Title: Bedside Ultrasound on the Effectiveness of Lumbar Puncture in Children - Open-label Randomized Trial
Brief Title: Bedside Ultrasound on the Effectiveness of Lumbar Puncture in Children.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KB/278/2023
Record Dates: First submitted 2024-08-02; First posted 2024-09-05 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Meningitis; Pediatric Disorder
MeSH Terms: conditions — Meningitis

STUDY DESIGN:
Intervention Model Description: Open-label, randomized interventional study
Masking Description: open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Utrasound group (Experimental): Bedside ultrasound examination of the lumbar spinal canal before lumbar puncture
  Interventions: Diagnostic Test: bedside ultrasound examination of the lumbar spinal canal
- Standard group (No Intervention): Standard procedure group

INTERVENTIONS:
Diagnostic Test: bedside ultrasound examination of the lumbar spinal canal — The ultrasound examination will be performed using a Lumify linear probe (frequency range 4-12 MHz). In the longitudinal projection, the doctor will assess the spinal cord endings by marking them with a sterile marker - a horizontal line on the patient's back. In the same projection, the doctor will designate a safe and optimal place (the greatest width of the dural sac) for performing a lumbar puncture by marking it with a sterile marker. Additionally, in the longitudinal projection, the researcher will measure the depth from the skin surface to the dura mater. Then, in the transverse projection, the doctor will confirm the absence of the spinal cord at the planned puncture site and the optimal amount of cerebrospinal fluid in the selected space. This information will be passed on to the operator, who will ultimately decide on the lumbar puncture site.
  Arms: Utrasound group

SUMMARY:
The aim of the study is to assess the influence of ultrasound examination of the lumbar spinal canal on the effectiveness of lumbar puncture. An open-label, randomized interventional study.

DETAILED DESCRIPTION:
Lumbar puncture is a common procedure performed in pediatric departments. The most common purpose of the examination in the pediatric patient population is to exclude infectious diseases of the central nervous system: meningitis and encephalitis. Risk factors for traumatic or unsuccessful puncture include, among others: patient age less than 3 months, difficulty in identifying anatomical structures by palpation, lack of local anesthesia, lack of experience of the person performing the procedure, and patient movement during puncture. The use of spinal canal ultrasonography before performing lumbar puncture brings promising benefits. Ultrasound imaging can be helpful in visualizing key anatomical structures within the spinal canal and increasing the certainty of correct performance of the procedure, especially in inexperienced physicians.

The study objective is to assess the effect of ultrasound imaging of the lumbar spinal canal on the effectiveness of lumbar puncture.

We plan to include every child <18 years old with an indication for lumbar puncture to the one of the two groups (ultrasound group and standard group)

Before the procedure, doctors performing the lumbar puncture in both groups will complete a questionnaire regarding their previous experience In the USG group, before performing the lumbar puncture, one of the two researchers will perform a bedside ultrasound examination of the lumbar spinal canal.

The ultrasound examination will be performed using a Lumify linear probe (frequency range 4-12 MHz). In the longitudinal projection, the doctor will assess the sites of the spinal cord endings by marking them with a sterile marker - a horizontal line on the patient's back. In the same projection, the doctor will designate a safe and optimal site (the greatest width of the dural sac) for performing a lumbar puncture by marking it with a sterile marker. Additionally, in the longitudinal projection, the researcher will measure the depth from the skin surface to the dura mater. Then, in the transverse projection, the doctor will confirm the absence of the spinal cord at the planned puncture site and the optimal amount of cerebrospinal fluid in the selected space. This information will be passed on to the operator, who will ultimately decide on the location of the lumbar puncture.

In patients in the control group, the lumbar puncture will be performed by palpation, without additional interventions. The position of the patient in both groups will depend on the preferences of the physician performing the puncture. The procedure time will be measured from the moment the needle pierces the skin until the moment of obtaining cerebrospinal fluid or removing the needle if the fluid is not obtained. In the research group, the time of the ultrasound examination will be additionally measured.

ELIGIBILITY:
Inclusion Criteria:

* children <18 years of age
* patients who are scheduled to undergo lumbar puncture
* consent of legal guardian

Exclusion Criteria:

* infection of skin and tissues in the area of planned puncture
* developmental defects of the spine and spinal cord
* lack of consent of legal guardian
* contraindications to lumbar puncture

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Obtaining cerebrospinal fluid after the first attempt at lumbar puncture | 1 day
  Obtaining cerebrospinal fluid after the first attempt at lumbar puncture (at least 0.5 ml in volume, with a red blood cell count of <10,000/mm3).

SECONDARY OUTCOMES:
obtaining cerebrospinal fluid - < 10,000/mm3 - at any attempt | 1 day
  obtaining cerebrospinal fluid (volume min. 0.5 ml, with erythrocyte count < 10,000/mm3) in subsequent puncture attempts
obtaining cerebrospinal fluid - > 10,000/mm3 - at any attempt | 1 day
  obtaining bloody cerebrospinal fluid (volume min. 0.5 ml, with erythrocyte count > 10,000/mm3)
total number of puncture attempts to obtain cerebrospinal fluid | 1 day
  total number of puncture attempts to obtain cerebrospinal fluid in each patient (next puncture will be understood as another puncture of the skin with a needle)
unsuccessful puncture - failure to obtain cerebrospinal fluid | 1 day
  total number of participants with unsuccessful puncture - failure to obtain cerebrospinal fluid
duration of puncture | 1 day
  Mean duration of puncture for each patient Measured from the moment of puncturing the skin with the needle to the moment of obtaining cerebrospinal fluid or removal of the needle in the case of unsuccessful puncture.
  Measured in seconds.
assessment of the impact of ultrasound imaging on the effectiveness of lumbar puncture depending on the experience of the physician performing the lumbar puncture | 1 day
  Difference in success rate depending on experience - measured by the number of punctures performed so far) puncture: 0-5 low experience, 6-15 medium experience, >15 high experience.
assessment of the impact of ultrasound imaging on the effectiveness of lumbar puncture depending on the patient's BMI z-score | 1 day
  Difference in success rate depending onthe patient's BMI z-score

CONTACTS AND LOCATIONS:
Overall Officials: Agata Ćwiek, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Medcial Univeristy of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided